CLINICAL TRIAL: NCT02307864
Title: A Randomized, Double-Blind, Placebo- and Positive-Controlled, Multiple Dose, Four Way Crossover Study to Evaluate the Effects of Tramadol Hydrochloride on Cardiac Repolarization in Healthy Subjects at Therapeutic and Supratherapeutic Dose Levels
Brief Title: Study to Evaluate the Effects of Tramadol Hydrochloride on Cardiac Repolarization in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Collaborators: Bausch Health Americas, Inc. (Industry); Cipher Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CR106355; TRAMPAI1003 (Other: Janssen Scientific Affairs, LLC); V01-TRAA-401 (Other: Valeant Pharmaceuticals International Inc); 2014-01-00 (Other: Cipher Pharmaceuticals Inc)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: Healthy; QT interval; QTc interval; Electrocardiogram; Tramadol hydrochloride; Moxifloxacin; Placebo
MeSH Terms: interventions — Tramadol; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- Treatment Sequence 1 (Experimental): Participants will receive treatment A (2*50 milligram [mg] tramadol hydrochloride [HCl] immediate release [IR] tablet + 1 tramadol HCl placebo every 6 hours on Days 1, 2, and 3, along with single dose of 2*50 mg tramadol HCl IR tablet + 1 tramadol HCl placebo + 1 moxifloxacin placebo on Day 4); treatment B (3*50 mg tramadol HCl IR tablet every 6 hours on Days 1, 2, and 3, along with single dose of 3*50 mg tramadol HCl IR tablet + 1 moxifloxacin placebo on Day 4); treatment C (3 tramadol HCl placebo every 6 hours on Days 1, 2, and 3, along with single dose of 3 tramadol HCl placebo + 1 moxifloxacin placebo on Day 4); and treatment D (3 tramadol HCl placebo every 6 hours on Days 1, 2, and 3, along with single dose of 3 tramadol HCl placebo + 1 moxifloxacin placebo on Day 4) in 4 treatment periods as per protocol defined sequence. A washout period of 7 to 15 days will be maintained between each treatment period.
  Interventions: Drug: Tramadol HCl; Drug: Moxifloxacin 400 mg; Drug: Tramadol HCl Placebo; Drug: Moxifloxacin Placebo
- Treatment Sequence 2 (Experimental): Participants will receive treatment A; treatment B; treatment C; and treatment D in 4 treatment periods as per protocol defined sequence. A washout period of 7 to 15 days will be maintained between each treatment period.
  Interventions: Drug: Tramadol HCl; Drug: Moxifloxacin 400 mg; Drug: Tramadol HCl Placebo; Drug: Moxifloxacin Placebo
- Treatment Sequence 3 (Experimental): Participants will receive treatment A; treatment B; treatment C; and treatment D in 4 treatment periods as per protocol defined sequence. A washout period of 7 to 15 days will be maintained between each treatment period.
  Interventions: Drug: Tramadol HCl; Drug: Moxifloxacin 400 mg; Drug: Tramadol HCl Placebo; Drug: Moxifloxacin Placebo
- Treatment Sequence 4 (Experimental): Participants will receive treatment A; treatment B; treatment C; and treatment D in 4 treatment periods as per protocol defined sequence. A washout period of 7 to 15 days will be maintained between each treatment period.
  Interventions: Drug: Tramadol HCl; Drug: Moxifloxacin 400 mg; Drug: Tramadol HCl Placebo; Drug: Moxifloxacin Placebo

INTERVENTIONS:
Drug: Tramadol HCl — Tramadol HCl 50 mg immediate release (IR) tablet administered orally.
  Other Names: RWJ-26898-002
Drug: Moxifloxacin 400 mg — Moxifloxacin 400 mg tablet administered orally.
  Other Names: Avelox
Drug: Tramadol HCl Placebo — Placebo matched to tramadol HCl IR tablet administered orally.
Drug: Moxifloxacin Placebo — Placebo matched to Moxifloxacin 400 mg tablet administered orally.

SUMMARY:
The purpose of this study is to assess the effects of multiple doses of an immediate release (IR) formulation of tramadol hydrochloride (HCl) at therapeutic and supratherapeutic levels in healthy adult participants on the electrocardiogram (ECG) QT interval corrected for heart rate (QTc).

DETAILED DESCRIPTION:
This is a randomized (study medication assigned by chance), double-blind (neither physician nor participant knows the treatment that the participant receives), 4-way crossover (method used to switch participants from one treatment arm to another), placebo- and positive-controlled (the experimental treatment or procedure is compared to an inactive substance and a standard treatment or procedure), single site, multiple dose study. The study has 3 phases: a Screening Phase (up to 35 days); a Double-blind Treatment Phase (4 treatment periods with a washout period of 7 to 15 days); and a Post-treatment Phase (Day 5 of Period 4 or at the time of early withdrawal). All eligible participants will receive each of the 4 treatments: tramadol HCl at therapeutic dose of 400 milligram per day (mg/day), tramadol HCl at supratherapeutic dose of 600 mg/day, placebo, and positive control moxifloxacin 400 mg; in any of the treatment period as per assigned treatment sequence. The total duration of each participant's participation will be up to a maximum of 100 days. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Woman participant of child-bearing potential, must have a negative serum beta-human chorionic gonadotropin pregnancy test at Screening; and a negative urine pregnancy test on Day 1 of each treatment period
* Standard electroencephalogram (EEG) that is normal, as assessed by a neurologist. The EEG will be performed under basic conditions and during hyperventilation and intermittent photic stimulation at Screening
* Body mass index (BMI; weight [in kilogram]/height [in square meter]) between 18 and 30 kilogram per square meter (inclusive), and body weight not less than 50 kilogram at Screening
* Blood pressure between 90 and 140 millimeter of mercury (mm Hg) systolic (inclusive) and no higher than 90 mm Hg diastolic
* An average of triplicate 12-lead electrocardiogram (ECG) recordings (performed in a semi-supine position), completed within 4 minutes total, consistent with normal cardiac conduction and function at Screening, including: 1- Sinus rhythm with heart rate between 40 and 100 beats per minute (inclusive); 2- QTc interval between 350 to 450 milliseconds (inclusive); 3- QRS interval of less than 110 milliseconds; 4- PR interval less than 200 milliseconds; 5- ECG morphology consistent with healthy cardiac conduction and function

Exclusion Criteria:

* Personal or family history of epileptic seizures or convulsions (genetic or idiopathic seizures), or have suffered from head trauma with loss of consciousness, central nervous system infection, or loss of consciousness of unknown origin
* History of additional risk factors for torsades de pointes (TdP) or the presence of a family history of short QT syndrome, long QT syndrome, sudden unexplained death at a young age ( less than equal to 40 years), drowning or sudden infant death syndrome in a first degree relative (that is, biological parent, sibling, or child)
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at Screening or before the first dose of study drug on Day -1 of each treatment period as assessed by the Investigator. Note that participants who have serum potassium, magnesium, or calcium levels outside of the local laboratory's reference range will be excluded
* Clinically significant abnormal physical examination or vital signs at Screening or before the first dose of study drug on Day -1 of each treatment period as assessed by the Investigator
* History of drug or alcohol abuse within 5 years before Screening or positive test result(s) for alcohol or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines, hallucinogens, and benzodiazepines) at Screening or on Day -1 of each treatment period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2015-08-22 (Actual); Study Completion 2015-08-27 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in QTc Interval | Baseline (pre-dose, Day1); pre-dose up to 24 hours post-dose on Day 4
  The QT interval corrected for heart rate (QTc interval) using Fridericia, Bazett and study-specific power correction methods, will be measured by electrocardiograms (ECG).

SECONDARY OUTCOMES:
Change From Baseline in HR, QRS, and PR Intervals | Baseline (pre-dose, Day1); pre-dose up to 24 hours post-dose on Day 4
  The HR, QRS, and PR Intervals, will be measured by ECG.
Number of Participants with T-wave and U-wave Morphological Changes | Baseline (pre-dose, Day1); pre-dose up to 24 hours post-dose on Day 4
  The number of participants having T wave morphology changes from baseline and/or the occurrence of abnormal U-waves that represent the appearance or worsening of the morphological abnormality will be reported.
Maximum Plasma Concentration During a Dosing Interval at Steady State (Cmax,ss) | Pre-dose up to 24 hours post-dose on Day 4
  The Cmax,ss is the maximum plasma concentration at steady state which will be observed during a dosing interval.
Trough Plasma Concentration Before Dosing (pre-dose) At Steady State (Ctrough,ss) | Pre-dose up to 24 hours post-dose on Day 4
  The Ctrough,ss refers to the drug concentration at steady state, at the time when it is expected to reach its minimum (trough) concentration.
Time to Reach the Maximum Plasma Concentration at Steady State (Tmax,ss) | Pre-dose up to 24 hours post-dose on Day 4
  The Tmax,ss is the time to reach maximum plasma concentration at steady state which will be observed during a dosing interval.
Area Under the Plasma Concentration-Time Curve During a Dosing Interval (tau) at Steady State (AUCtau,ss) | Pre-dose up to 24 hours post-dose on Day 4
  The AUC (tau,ss) is the area under the plasma concentration time curve observed during a dosing interval (tau) at steady state.
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Screening up to end of study (30 days after the last dose of study drug or early withdrawal)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (1):
- Overland Park, Kansas, United States